CLINICAL TRIAL: NCT06016426
Title: Mass Closure vs Layer by Layer Closure of the Transverse Abdominal Laparotomy Incisions in Infants and Children: a Randomized Clinical Trial
Brief Title: Mass Closure vs Layer by Layer Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammad Gharieb Mohammad Khirallah, professor of pediatric surgery, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 36264PR286/8/23
Record Dates: First submitted 2023-08-18; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Abdominal Wall Wound; Ventral Hernia; Incisional Hernia
Keywords: transverse laparotomy; incisional hernia; mass closure; layer by layer closure
MeSH Terms: conditions — Hernia, Ventral; Incisional Hernia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mass closure (Active Comparator): infants and children whose transverse laparotomy incisions will be closed in mass closure.
  Interventions: Other: Mass closure vs layer by layer closure of transverse laparotomy incisions in children and infants.
- layer by layer closure (Active Comparator): infants and children whose transverse laparotomy incisions will be closed layer by layer.
  Interventions: Other: Mass closure vs layer by layer closure of transverse laparotomy incisions in children and infants.

INTERVENTIONS:
Other: Mass closure vs layer by layer closure of transverse laparotomy incisions in children and infants. — the transverse laparotomy incision in infants and children will be either closed as single layer included the peritoneum, posterior rectus sheath and anterior rectus sheath wit muscle sparing, or the laparotomy will be closed in layer by layer in which the peritoneum and posterior rectus sheath are closed as a layer and the anterior rectus sheath is closed as a seprate layer.

SUMMARY:
to assess two different ways of closure of laparotomy in children and infants

DETAILED DESCRIPTION:
Introduction:

The technique of abdominal wall closure in infants subjected to abdominal transverse laparotomy incision may have an impact not only on the development of a future incisional hernia but also on the function of the anterior abdominal wall muscles.

There are two ways to close this laparotomy incision. These ways are either closure in mass or layer by layer closure. Neither of them is superior to the other.

The main issue that minds the pediatric surgeons is a safe and successful repair of the abdominal wall incision and the avoidance of the development of incisional hernia.

The aim of this work is to randomly compare the two different techniques of the closure of transverse laparotomy incision.

Patients and methods:

- Study design: The study was performed during the period from January 2020 to October 2024. It is a randomized control trial.

Inclusion criteria were infants younger than 3 years. We excluded infants with history of prematurity, previous abdominal operations and infants with congenital abdominal wall defects.

An informed consent was obtained from the parents or the care giver of every participant.

Randomization was obtained using closed envelop method. Patients were categorized into two groups A and B. Group A included patients that their exploratory wound was closed with mass closure method using Vicryl® 2/0 round needle. Group B included patients that their exploratory wound was closed layer by layer using the same suture material.

In both groups the ratio of the suture length to the wound was 3 to 1. - The measured variables: The variables that were addressed were

1. the mean operative time in minutes,
2. the incidence of wound dehiscence,
3. the occurrence of wound infection,
4. The development of an incisional hernia
5. Long term assessment of both abdominal wall structure and dynamics of abdominal muscles at the site of incision.

   * Follow up protocol:

All patients were scheduled on a follow up regimen. They were examined weekly for one month post-operative. Then monthly for one year. The anterior abdominal wall of these patients was examined by ultrasound at the 6th and 12th moth postoperatively. This helped assessment of the dynamics and structure of the muscles at the site of the incision.

- Statistical analysis: Statistical analysis was conducted using SPSS ™ statistical package ver. 21 (IBM SPSS, NY, USA). Numerical data were compared using an independent sample t-test, whereas categorical data were compared using the chi-square test. Statistical significance was set at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* all infants and children with transverse laparotomy

Exclusion Criteria:

* previous abdominal operations
* children and infants with congenital abdominal wall defects

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
wound failure with the development of incisional hernia later in either group | one year
  the occurrence or development of the incisional hernia is the primary outcome. the incidence of the development of this hernia will be recorded in each group. this will help choose the more appropriate method of transverse laparotomy closure in infants and children

SECONDARY OUTCOMES:
surgical site infections | two weeks up to one month
  the number of patients who will develop a surgical site infections in each group, the mean duration of hospital stay if this happened. the number of patients who will later develop an incisional hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided